CLINICAL TRIAL: NCT06064396
Title: Effects of Gong's Mobilization With and Without Stecco Fascial Therapy in Patients With Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0136 Ifra Awan
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive Capsulitis; Pain; Range of Motion
MeSH Terms: conditions — Bursitis; Pain

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of the treatment arms at the beginning of the trial and continue in that arm throughout the length of the trial.
Who Masked: Outcomes Assessor
Masking Description: Blinding,refers to a practice where study participants are prevented from knowing certain information that may somehow influence them-thereby tainting the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gong's Mobilization with Stecco Fascial Therapy (Experimental): Participants in this group will receive Gong's Mobilization with Stecco Fascial Therapy
  Interventions: Other: Gong's Mobilization; Other: Stecco Fascial Therapy
- Gong's Mobilization (Active Comparator): Participants in this group will receive Gong's Mobilization
  Interventions: Other: Gong's Mobilization

INTERVENTIONS:
Other: Gong's Mobilization — The duration of intervention will be 4 weeks, 3 sessions a week, a total of 12 sessions will be given to the study participants. Each session will last for 30 minutes. Conventional physical therapy will be given to participants along with Gong's Mobilization.
Other: Stecco Fascial Therapy — The duration of intervention will be 4 weeks, 3 sessions a week, a total of 12 sessions will be given to the study participants. Each session will last for 30 minutes. Conventional physical therapy will be given to participants along with stecco fascial therapy.
  Arms: Gong's Mobilization with Stecco Fascial Therapy

SUMMARY:
The aim of this study is to determine the effects of Gong's mobilization with and without Stecco Fascial therapy on pain, range of motion and function in patients with Adhesive capsulitis.

DETAILED DESCRIPTION:
Adhesive capsulitis is characterized by a painful, progressive loss of both active and passive glenohumeral mobility that results from the glenohumeral joint capsule's increasing fibrosis and eventual rigidity. The clinical syndrome known as "frozen shoulder" restricts active and passive range of motion (ROM) in flexion, abduction, and rotation, among other movements.

A research conducted on effectiveness of Gong's mobilisation versus muscle energy technique on pain and functional ability of shoulder in phase II adhesive capsulitis. He included 50 subjects and then randomly allocated them into two groups. Duration of treatment was 6 sessions per week for two weeks. The Gong's mobilisation (Group A) pull was maintained for about 10-15 seconds. Maitland's grade 3 and 4 was performed to increase the range. Muscle energy technique was applied for 5 repetitions per set, 5 days a week for 2 weeks. Group A showed significant improvement than Group B. This implies that Gong's mobilisation is more beneficial in improving ROM, reducing pain, improving functional ability.

A study conducted to determine the effect of Fascial Manipulation on the Internal Rotation Range of Motion in athletes with GIRD. Asymptomatic overhead athletes with GIRD more than 20° when compared with the non-dominant shoulder were randomly assigned to two groups. The experimental group has received three sessions of FM treatment in two weeks. FM applied to densified Centre of Coordination (CC) points located on the myofascial sequences for 5 to 8 minutes at each CC point. The control group has received three sessions of posterior shoulder capsule release using a tennis ball under supervision.This study indicates that FM may be used as an adjunct to stretching in asymptomatic participants with GIRD to increase the IRROM.

There is limited literature available regarding the combined effects of Gong's Mobilization with Stecco Fascial manipulative therapy on pain, range of motion and function in patients with adhesive capsulitis. Previous literature was carried on smaller sample size and for two weeks without any follow up. In previous studies long term effects were not known and only shoulder abduction and internal rotation range of motion were measured. Therefore, in this study combined effects of Gong's mobilization and Stecco Fascial Therapy will be study on pain, range of motion and function in patients with Adhesive Capsulitis. This study will include all range of motion of shoulder joint and also include home plan after the session.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients
* Patients with positive capsular pattern of glenohumeral joint which is external rotation, abduction and internal rotation
* Patients aged 35-60 years with shoulder pain and reduction in range of motion
* Unilateral stage II frozen shoulder with shoulder pain and stiffness for more than 3 months

Exclusion Criteria:

* Patients with additional cervical or shoulder pathology
* Patients with shoulder dislocation, rotator cuff rupture and injury
* Medical red flag history (tumor, metabolic diseases, rheumatoid arthritis, osteoporosis or Infection)
* Neurological disorder or symptomatic herniated disc or severe disorders of the cervical spine
* History of Severe trauma or any fracture or surgery

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Pain: Numeric Pain Rating Scale (NPRS) | 4th week
  Changes from baseline Numeric pain rating scale is The 11-point scale used to capture the patient's level of pain. The scale is anchored on the left with the phrase ''no pain'' and on the right with the phrase ''worst imaginable pain.'' Patients rate their current level of pain and their worst and least amount of pain in the last 24 hours. Numeric pain scales have been shown to be reliable and valid with validity range from 0.86 to 0.95 and high test-retest reliability r=0.96
Range of Motion Shoulder (Flexion) | 4th week
  Changes from baseline ROM range of motion of shoulder flexion will be taken with the help of universal goniometer.
Range of Motion Shoulder (Abduction) | 4th week
  Changes from baseline ROM range of motion of shoulder abduction will be taken with the help of universal goniometer.
Range of Motion Shoulder (External rotation) | 4th week
  Changes from baseline ROM range of motion of shoulder external rotation will be taken with the help of universal goniometer.
Range of Motion Shoulder (Internal rotation) | 4th week
  Changes from baseline ROM range of motion of shoulder internal rotation will be taken with the help of universal goniometer.
Function: Shoulder Pain and Disability Index (SPADI) Questionnaire | 4th week
  Changes from baseline SPADI. SPADI questionnaire is used for the self-assessment of symptoms and function of the shoulder. 13 items (total score): 5 items for pain and 8 for function (sub scores). Response options/scale. All SPADI items are originally scored on a visual analog scale (VAS) from no pain/no difficulty to worst pain imaginable/so difficult required help. The VAS line was divided into 12 equal intervals to obtain a 12-point numerical rating scale (NRS) ranging from 0 (best) to 11 (worst).

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, Phd, Principal Investigator — Riphah International University
Locations (1):
- Arif Memorial Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neviaser AS, Hannafin JA. Adhesive capsulitis: a review of current treatment. Am J Sports Med. 2010 Nov;38(11):2346-56. doi: 10.1177/0363546509348048. Epub 2010 Jan 28. PMID 20110457
- [Background] Tasto JP, Elias DW. Adhesive capsulitis. Sports Med Arthrosc Rev. 2007 Dec;15(4):216-21. doi: 10.1097/JSA.0b013e3181595c22. PMID 18004221
- [Background] Wang K, Ho V, Hunter-Smith DJ, Beh PS, Smith KM, Weber AB. Risk factors in idiopathic adhesive capsulitis: a case control study. J Shoulder Elbow Surg. 2013 Jul;22(7):e24-9. doi: 10.1016/j.jse.2012.10.049. Epub 2013 Jan 24. PMID 23352186
- [Background] Tighe CB, Oakley WS Jr. The prevalence of a diabetic condition and adhesive capsulitis of the shoulder. South Med J. 2008 Jun;101(6):591-5. doi: 10.1097/SMJ.0b013e3181705d39. PMID 18475240
- [Background] Wadsworth CT. Frozen shoulder. Phys Ther. 1986 Dec;66(12):1878-83. doi: 10.1093/ptj/66.12.1878. PMID 3786418
- [Background] Celik D. Comparison of the outcomes of two different exercise programs on frozen shoulder. Acta Orthop Traumatol Turc. 2010;44(4):285-92. doi: 10.3944/AOTT.2010.2367. PMID 21252605
- [Background] Day JA, Stecco C, Stecco A. Application of Fascial Manipulation technique in chronic shoulder pain--anatomical basis and clinical implications. J Bodyw Mov Ther. 2009 Apr;13(2):128-35. doi: 10.1016/j.jbmt.2008.04.044. Epub 2008 Jun 24. PMID 19329049
- [Background] Russell S, Jariwala A, Conlon R, Selfe J, Richards J, Walton M. A blinded, randomized, controlled trial assessing conservative management strategies for frozen shoulder. J Shoulder Elbow Surg. 2014 Apr;23(4):500-7. doi: 10.1016/j.jse.2013.12.026. PMID 24630545